CLINICAL TRIAL: NCT01167777
Title: Multi-center Evaluation of the VERSANT® CT/GC DNA 1.0 Assay (kPCR)in Detecting C. Trachomatis and N. Gonorrhoeae
Status: Terminated | Type: Observational
Why Stopped: Siemens Management decided not to release the product in the USA.
Sponsor: Siemens Healthcare Diagnostics Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: MCSA-VkPCRCTGC-200810-PRO
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Chlamydia; Gonorrhea
Keywords: CT; GC; NG; chlamydia; gonorrhoeae
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- male/female: Symtomatic and asymptomatic males and females attending STD, family planning, public health and women's health clinics, or other applicable centers, who are being screened for CT or GC.

SUMMARY:
Multicenter clinical study to test a new qualitative in vitro nucleic acid amplification assay based on kPCR technology. The assay is intended for the diagnosis of Chlamydia trachomatis (CT) and Neisseria gonorrhoeae (GC).

DETAILED DESCRIPTION:
The study was terminated

This clinical trial protocol outlines the analytical and clinical performance characteristics that will be evaluated to demonstrate equivalency of the VERSANT CT/GC DNA 1.0 (kPCR) Assay for product registration. The Gen-Probe APTIMA Combo 2 Assay will be used as the CE-marked comparative method. The studies conducted during the clinical trial are intended to provide data to support the safety and effectiveness, as well as the labeling claims for the VERSANT CT/GC Assay. The study objectives are as follows:

* To demonstrate concordance with the Gen-Probe APTIMA Combo 2 Assay;
* To estimate the positive and negative predictive values for each specimen type included in the study;
* To estimate the indeterminate rate for each specimen type included in the study;
* To estimate the equivocal rate for each specimen type; and
* To assess reproducibility of the VERSANT CT/CG DNA 1.0 Assay (kPCR) using the VERSANT kPCR Molecular System.

Two (2) studies will be conducted to validate the analytical and clinical performance characteristics of the CT/GC DNA 1.0 (kPCR) Assay. Table 1 provides an overview of these studies.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older.
* Subject signed an IRB approved informed consent form.
* Subject is able to follow verbal and written instructions.

Exclusion Criteria:

* Subject has been on antibiotic therapy within 21 days prior to study enrollment.
* Subject urinated within one hour prior to sample collection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic and asymptomatic male and female patients attending STD, family planning, public health and women's health clinics, or other applicable centers, who are being screened for CT or GC
Sampling Method: Non-Probability Sample
Enrollment: 2296 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of CT and/or GC disease by clinical site | Study terminated

CONTACTS AND LOCATIONS:
Overall Officials: NORMAND DESPRES, PhD, Study Director — Siemens Healthcare Diagnostics
Locations (7):
- United States (7):
  - University of Alabama At Birmingham, Birmingham, Alabama
  - Los Angeles County Department of Public Health, Los Angeles, California
  - San Francisco Dept of Public Health, San Francisco, California
  - San Joaquin County Public Health Services, Stockton, California
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Hennepin County Medical Center, Minneapolis, Minnesota